CLINICAL TRIAL: NCT01431014
Title: The Effect of Steroid on Reducing Facial Swelling After Orthognathic Surgery
Brief Title: Effect of Steroid for the Postoperative Swelling After Orthognathic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 99-2811-B-182A-003; CGMH-IRB-100-2191B (Registry Identifier: CGMH IRB)
Record Dates: First submitted 2011-08-28; First posted 2011-09-09 (Estimated); Results first posted 2014-03-21 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2011-09

CONDITIONS: Swelling
Keywords: orthognathic surgery; steroid; swelling; 3-dimensional photogrammetry

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone"low-dose" (Active Comparator): 5mg
  Interventions: Drug: Dexamethasone"low-dose"
- Dexamethasone"high-dose" (Experimental): 15mg
  Interventions: Drug: Dexamethasone"high-dose"

INTERVENTIONS:
Drug: Dexamethasone"low-dose" — 5mg
  Other Names: dexan
  Arms: Dexamethasone"low-dose"
Drug: Dexamethasone"high-dose" — 15 mg
  Other Names: dexan
  Arms: Dexamethasone"high-dose"

SUMMARY:
Postoperative swelling is one of most common concerns to plastic and oromaxillary surgeons after orthognathic surgery. The purpose of this study is to develop a steroid regimen protocol for minimizing postoperative facial swelling after orthognathic surgery.

DETAILED DESCRIPTION:
Postoperative swelling is an annoying problem after orthognathic surgery. There are two reasons to minimize postoperative swelling. The first is a functional consideration. Orthognathic surgery is performed in oromaxillary area, and consequently swelling in this area can compromise airway. The second is esthetic one, as patients feel uncomfortable and embarrassing with a swollen face. Reducing facial swelling after orthognathic surgery helps to reduce airway complication and patient down time.

Several methods are used to reduce postoperative facial swelling, including controlled hypotension during operation, meticulous operative procedures, postoperative facial ice packing, head elevation, and suction drainage. Perioperative use of steroid has been applied for reduction of facial swelling after oral surgery and 3rd molar extraction. Cyclooxygenase-1 (COX1) and COX2 have been reported to be important enzymes for inflammatory process, and steroids inhibit their synthesis, consequently reducing postoperative edema. Steroid has also been used to decrease edema after orthognathic surgery, as well as to reduce pain, nausea and vomiting.

There were three randomized controlled studies looking at the effect of steroid on postoperative facial swelling after orthognathic surgery, separately by Dr. Weber et al, Peillon et al, and Munro et al. However, the results were controversial. The first two studies concluded that the steroid use could reduce facial swelling. The other one did not find significant difference between the experimental and control groups. Another limitation of the previous studies was that they all used two-dimensional or non-objective methods for evaluation of the amount of swelling, which could be less accurate. Three-dimensional photogrammetry has been introduced in recent years, and has obtained satisfactory results over the conventional methods. The investigators have experience of applying the device for facial surface study, and the accuracy has been validated in our imaging laboratory.

The purpose of this study is to determine the effect of steroid for reduction of postoperative facial swelling determined by three-dimensional photographic method. 3dMD face scanner will be used. The 3-dimensional method makes no harm to patients. Patients will be seated during scanning and thus reducing possible inconvenience. There is no radiation hazard with this method. The image acquisition time is 2 milliseconds or less, and therefore no concern of motion artifacts. The first part of this study is to get information about the swelling curve after orthognathic surgery. 3dMD face scanning will be performed 5 times postoperatively every 12 hours after 24 hours of operation. When the postoperative timing of maximal facial swelling is obtained, the investigators will proceed to perform the second part of study, and the number of facial scanning is reduced. The second part of study involves recruiting 70 patients with prognathism. The patients will be carefully screened and selected by craniofacial surgeons. The patients will take preoperative and postoperative 3dMD image scanning. The recovery course and clinical outcome will be monitored. 3dMD face image data analysis will be performed for quantitative comparisons between the experimental and control groups.

ELIGIBILITY:
Inclusion Criteria:

* patients who receive LeFort I osteotomy of maxilla and bilateral sagittal split osteotomy of mandible

Exclusion Criteria:

* patients with local or systemic diseases
* patients taking aspirin, steroid, nonsteroidal anti-inflammatory drugs, or having contraindications for steroids
* patients with history of psychosis
* patients with active or chronic infection
* patients with active or latent peptic ulcer

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lun-Jou Lo, MD, Principal Investigator — Chang Gung Memorial Hospital; Hye-Young Kim, MD, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan, Taiwan

REFERENCES:
- [Result] Kau CH, Cronin AJ, Richmond S. A three-dimensional evaluation of postoperative swelling following orthognathic surgery at 6 months. Plast Reconstr Surg. 2007 Jun;119(7):2192-2199. doi: 10.1097/01.prs.0000260707.99001.79. PMID 17519721
- [Result] van Loon B, Maal TJ, Plooij JM, Ingels KJ, Borstlap WA, Kuijpers-Jagtman AM, Spauwen PH, Berge SJ. 3D Stereophotogrammetric assessment of pre- and postoperative volumetric changes in the cleft lip and palate nose. Int J Oral Maxillofac Surg. 2010 Jun;39(6):534-40. doi: 10.1016/j.ijom.2010.03.022. Epub 2010 Apr 27. PMID 20427150
- [Result] Schaberg SJ, Stuller CB, Edwards SM. Effect of methylprednisolone on swelling after orthognathic surgery. J Oral Maxillofac Surg. 1984 Jun;42(6):356-61. doi: 10.1016/s0278-2391(84)80006-3. PMID 6585512
- [Result] Meyer-Marcotty P, Alpers GW, Gerdes AB, Stellzig-Eisenhauer A. Impact of facial asymmetry in visual perception: a 3-dimensional data analysis. Am J Orthod Dentofacial Orthop. 2010 Feb;137(2):168.e1-8; discussion 168-9. doi: 10.1016/j.ajodo.2008.11.023. PMID 20152669
- [Result] Rana M, Gellrich NC, Joos U, Piffko J, Kater W. 3D evaluation of postoperative swelling using two different cooling methods following orthognathic surgery: a randomised observer blind prospective pilot study. Int J Oral Maxillofac Surg. 2011 Jul;40(7):690-6. doi: 10.1016/j.ijom.2011.02.015. Epub 2011 Mar 15. PMID 21411291
- [Result] Chegini S, Dhariwal DK. Review of evidence for the use of steroids in orthognathic surgery. Br J Oral Maxillofac Surg. 2012 Mar;50(2):97-101. doi: 10.1016/j.bjoms.2010.11.019. Epub 2011 Feb 12. PMID 21316821
- [Result] Dan AE, Thygesen TH, Pinholt EM. Corticosteroid administration in oral and orthognathic surgery: a systematic review of the literature and meta-analysis. J Oral Maxillofac Surg. 2010 Sep;68(9):2207-20. doi: 10.1016/j.joms.2010.04.019. Epub 2010 Jun 29. PMID 20591548
- [Result] Bourke DL. Use of steroids during orthognathic surgery. J Oral Maxillofac Surg. 1986 Jan;44(1):2-3. doi: 10.1016/0278-2391(86)90004-2. No abstract available. PMID 3455720
- [Result] Weber CR, Griffin JM. Evaluation of dexamethasone for reducing postoperative edema and inflammatory response after orthognathic surgery. J Oral Maxillofac Surg. 1994 Jan;52(1):35-9. doi: 10.1016/0278-2391(94)90010-8. PMID 8263640
- [Result] Mocan A, Kisnisci R, Ucok C. Stereophotogrammetric and clinical evaluation of morbidity after removal of lower third molars by two different surgical techniques. J Oral Maxillofac Surg. 1996 Feb;54(2):171-5. doi: 10.1016/s0278-2391(96)90441-3. PMID 8604065
- [Result] Esen E, Tasar F, Akhan O. Determination of the anti-inflammatory effects of methylprednisolone on the sequelae of third molar surgery. J Oral Maxillofac Surg. 1999 Oct;57(10):1201-6; discussion 1206-8. doi: 10.1016/s0278-2391(99)90486-x. PMID 10513866
- [Result] Seo K, Tanaka Y, Terumitsu M, Someya G. Efficacy of steroid treatment for sensory impairment after orthognathic surgery. J Oral Maxillofac Surg. 2004 Oct;62(10):1193-7. doi: 10.1016/j.joms.2004.06.033. PMID 15452804
- [Result] Day CJ, Robert T. Three-dimensional assessment of the facial soft tissue changes that occur postoperatively in orthognathic patients. World J Orthod. 2006 Spring;7(1):15-26. PMID 16548302
- [Result] Laureano Filho JR, Maurette PE, Allais M, Cotinho M, Fernandes C. Clinical comparative study of the effectiveness of two dosages of Dexamethasone to control postoperative swelling, trismus and pain after the surgical extraction of mandibular impacted third molars. Med Oral Patol Oral Cir Bucal. 2008 Feb 1;13(2):E129-32. PMID 18223530
- [Result] Huaman ET, Juvet LM, Nastri A, Denman WT, Kaban LB, Dodson TB. Changing patterns of hospital length of stay after orthognathic surgery. J Oral Maxillofac Surg. 2008 Mar;66(3):492-7. doi: 10.1016/j.joms.2007.08.025. PMID 18280382
- [Result] Meisami T, Musa M, Keller MA, Cooper R, Clokie CM, Sandor GK. Magnetic resonance imaging assessment of airway status after orthognathic surgery. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2007 Apr;103(4):458-63. doi: 10.1016/j.tripleo.2006.07.006. Epub 2006 Oct 27. PMID 17395062
- [Result] Sotto-Maior BS, Senna PM, de Souza Picorelli Assis NM. Corticosteroids or cyclooxygenase 2-selective inhibitor medication for the management of pain and swelling after third-molar surgery. J Craniofac Surg. 2011 Mar;22(2):758-62. doi: 10.1097/SCS.0b013e318207f3fe. PMID 21415660
- [Result] Daniels SE, Desjardins PJ, Bird SR, Smugar SS, Tershakovec AM. Rofecoxib 50 mg and valdecoxib 20 or 40 mg in adults and adolescents with postoperative pain after third molar extraction: results of two randomized, double-blind, placebo-controlled, single-dose studies. Clin Ther. 2006 Jul;28(7):1022-34. doi: 10.1016/j.clinthera.2006.07.005. PMID 16990080
- [Result] Fleming PS, Flood TR. Steroid-induced psychosis complicating orthognathic surgery: a case report. Br Dent J. 2005 Nov 26;199(10):647-8. doi: 10.1038/sj.bdj.4812929. PMID 16311560
- [Result] Galen DM, Beck M, Buchbinder D. Steroid psychosis after orthognathic surgery: a case report. J Oral Maxillofac Surg. 1997 Mar;55(3):294-7. doi: 10.1016/s0278-2391(97)90546-2. No abstract available. PMID 9054921
- [Result] Precious D, Armstrong J, Morrison A, Field C. The incidence of total hip replacement in orthognathic surgery patients receiving short-term steroid therapy. J Oral Maxillofac Surg. 1992 Sep;50(9):956-7. doi: 10.1016/0278-2391(92)90054-4. PMID 1506971

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexamethasone"High-dose": 15mg
  Dexamethasone"high-dose" : 15 mg
- Dexamethasone"Low-dose": 5mg
  Dexamethasone"low-dose" : 5mg
Period: Overall Study
Arm/Group | Dexamethasone"High-dose" | Dexamethasone"Low-dose"
Started | 34 | 34
Completed | 31 | 25
Not Completed | 3 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone"High-dose" | Dexamethasone"Low-dose" | Total
Number analyzed (Participants) | 31 | 25 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 5 | 6
  Between 18 and 65 years | 30 | 20 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.16 (4.19) | 20.92 (4.79) | 22.16 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 16 | 12 | 28
Region of Enrollment [Number; unit: participants]
  Taiwan | 31 | 25 | 56

OUTCOME MEASURES:

1. Primary Outcome: Effect of Perioperative Steroid for the Postoperative Swelling After Orthognathic Surgery
Description: Measure of facial swelling will be performed using 3-dimensional photogrammetry. The 3d photo acquisition is non-invasive without radiation concern. The images will be taken before and after surgery to measure and compare the degree of facial swelling. Side effects from the steroid use are expected to be low under normal clinical dosage, but will also be monitored. Symptoms of wound infection, psychosis, and prolonged wound healing will be studied. There should be no long term complication, since the steroid use is one single dose.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: ml
Groups:
- Dexamethasone"Low-dose": 5mg Dexamethasone"low-dose" : 5 mg
Arm/Group | Dexamethasone"High-dose" | Dexamethasone"Low-dose"
Number analyzed (Participants) | 31 | 25
ml
  36 hours postoperatively | 167.06 (55.93) | 190.73 (78.74)
  1week postoperatively | 61.39 (30.14) | 57.62 (36.13)
  1month postoperatively | 29.85 (19.40) | 19.34 (16.56)
Statistical Analysis 1: Comparison: Dexamethasone"High-dose" vs Dexamethasone"Low-dose"; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Dexamethasone"Low-dose" | Dexamethasone"High-dose"
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/31
Other Adverse Events (participants affected / at risk) | 0/25 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes